CLINICAL TRIAL: NCT02510079
Title: Emergent Expanded Access to Use Autologous Human Schwann Cell Augmentation of Nerve Autograft Repair in a Single Patient With Severe Peripheral Nerve Injury
Brief Title: Emergent Expanded Access for ahSC Augmentation of Nerve Autografts After Severe Peripheral Nerve Injury.
Status: No longer available | Type: Expanded Access
Sponsor: W. Dalton Dietrich (Other)
Collaborators: The Miami Project to Cure Paralysis (Other)
Responsible Party: Sponsor-Investigator, W. Dalton Dietrich, Professor of Neurosurgery, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20150501
Record Dates: First submitted 2015-07-15; First posted 2015-07-28 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Sciatic Nerve Injury

INTERVENTIONS:
Biological: Autologous human Schwann cells — Schwann cells harvested from the sural nerve will be autologously transplanted along sural nerve autografts wrapped in a collagen matrix (Duragen).

SUMMARY:
The primary purpose of this research study is to determine the safety of injecting ones own Schwann cells to augment sural nerve autografts after a severe, non-lacerating injury to the sciatic nerve has occurred.

DETAILED DESCRIPTION:
The secondary purpose of this research project is to evaluate whether transplanted Schwann cells can enhance recovery of sensory and motor function. Emergency expanded access for a single patient was granted, as the patient was an ideal candidate for sural nerve repair augmented by autologous Schwann cells which could be harvested from a relatively small segment of sensory nerve. The cells were expanded using cell culture techniques and placed along with the sural nerve grafts wrapped by an FDA approved collagen matrix (Duragen). This study is being conducted at the Jackson Memorial and the University of Miami health systems. As a research subject the patient will be in this study for a total of 5 years from the date receiving Schwann cell transplant augmentation of sural nerve autografts.

ELIGIBILITY:
Single patient with severe sciatic nerve injury enrolled under emergency request

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: W. Dalton Dietrich, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States